CLINICAL TRIAL: NCT00243633
Title: Characterization of Focal Liver Lesions by Real-time Contrast-enhanced Ultrasound Imaging (CEUS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIT 05 - FT / ECUS
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Focal Liver Lesions; Liver Cancer; Liver Cirrhosis
Keywords: focal liver lesions; contrast-enhanced ultrasound sonography; cirrhosis; suspected liver metastases; suspected liver cirrhosis
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Real-time contrast-enhanced ultrasound sonography

SUMMARY:
The conventional sonography is frequently used to detect incidental focal liver lesions because of its availability, innocuity and low cost. Nevertheless, sensibility and specificity of conventional sonography does not exceed 70% for tumoral affections. Consequently the interest of this practice must be reconsidered by studying its ratio cost/diagnosis contribution.

These limitations of conventional sonography have led to the use of other imaging modalities and invasive or costly procedures such as computed tomography (CT), magnetic resonance imaging (MRI) or biopsy. The availability of real-time contrast-enhanced ultrasound imaging (CEUS) has changed the strategy in the characterization of focal liver lesions, on healthy or cirrhotic liver in a neoplastic context or not, without inconvenience for the patient.

The aim of the present study is to evaluate the place of CEUS in term of diagnostic relevance and catch of load cost, in the characterization of focal liver lesions detected but not characterized by CT or conventional sonography.

ELIGIBILITY:
Inclusion Criteria:

* Target focal liver lesion of size lower than 10 cm and higher than 5 mm detected by conventional ultrasonography

Exclusion Criteria:

* Patients with acute coronary syndrome or clinically unstable ischaemic cardiac disease, including: myocardial infarction, recent coronary artery intervention, acute cardiac failure (within last month), acute endocarditis and prosthetic valves.
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Medical and economic interest of CEUS

SECONDARY OUTCOMES:
Method acceptability
Contrast-enhanced ultrasound sonography tolerance
Harmony inter-readers

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel CORREAS, Dr, Principal Investigator — Necker Hospital; François TRANQUART, Pr, Study Director — University Hospital, Tours
Locations (15):
- France (15):
  - CHRU d'ANGERS, Angers
  - Hôpital Saint-Jacques, CHRU Besancon, Besançon
  - Hôpital Saint-André, CHRU Bordeaux, Bordeaux
  - Hôpital Beaujon, Assistance Publique Hôpitaux de Paris, Clichy
  - Hospices Civils de Lyon, Lyon
  - Hôpital Saint-Eloi, CHRU Montpellier, Montpellier
  - Hôpital Pitié Salpétrière, Assistance Publique Hôpitaux de Paris, Paris
  - Hôpital Necker, Assistance Publique Hôpitaux de Paris, Paris
  - Hôpital La Milétrie, CHRU Poitiers, Poitiers
  - Hôpital Robert Debré, CHRU Reims, Reims
  - Hôpital Nord, CHRU Saint-Etienne, Saint-Etienne
  - Hôpital Bretonneau, CHRU Tours, Tours
  - Service de Radiologie, Hôpital d'Enfants de Brabois, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Assistance Publique Hôpitaux de Paris, Villejuif
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Kim TK, Choi BI, Hong HS, Choi BY, Han JK. Improved imaging of hepatic metastases with delayed pulse inversion harmonic imaging using a contrast agent SH U 508A: preliminary study. Ultrasound Med Biol. 2000 Nov;26(9):1439-44. doi: 10.1016/s0301-5629(00)00268-4. PMID 11179618
- [Background] Albrecht T, Blomley MJ, Burns PN, Wilson S, Harvey CJ, Leen E, Claudon M, Calliada F, Correas JM, LaFortune M, Campani R, Hoffmann CW, Cosgrove DO, LeFevre F. Improved detection of hepatic metastases with pulse-inversion US during the liver-specific phase of SHU 508A: multicenter study. Radiology. 2003 May;227(2):361-70. doi: 10.1148/radiol.2272011833. Epub 2003 Mar 20. PMID 12649417
- [Background] Quaia E, Bertolotto M, Forgacs B, Rimondini A, Locatelli M, Mucelli RP. Detection of liver metastases by pulse inversion harmonic imaging during Levovist late phase: comparison with conventional ultrasound and helical CT in 160 patients. Eur Radiol. 2003 Mar;13(3):475-83. doi: 10.1007/s00330-002-1670-1. Epub 2002 Sep 26. PMID 12594549
- [Background] Bernatik T, Becker D, Neureiter D, Hansler J, Frieser M, Schaber S, Hahn EG, Strobel D. [Detection of liver metastases--comparison of contrast--enhanced ultrasound using first versus second generation contrast agents]. Ultraschall Med. 2003 Jun;24(3):175-9. doi: 10.1055/s-2003-40060. German. PMID 12817311
- [Background] Basilico R, Blomley MJ, Harvey CJ, Filippone A, Heckemann RA, Eckersley RJ, Cosgrove DO. Which continuous US scanning mode is optimal for the detection of vascularity in liver lesions when enhanced with a second generation contrast agent? Eur J Radiol. 2002 Mar;41(3):184-91. doi: 10.1016/s0720-048x(01)00459-4. PMID 11861092
- [Background] Leen E, Angerson WJ, Yarmenitis S, Bongartz G, Blomley M, Del Maschio A, Summaria V, Maresca G, Pezzoli C, Llull JB. Multi-centre clinical study evaluating the efficacy of SonoVue (BR1), a new ultrasound contrast agent in Doppler investigation of focal hepatic lesions. Eur J Radiol. 2002 Mar;41(3):200-6. doi: 10.1016/s0720-048x(01)00457-0. PMID 11861094
- [Background] Tranquart F, Bleuzen A, Tchuenbou J. [Contrast ultrasound imaging in focal liver lesions: diagnostic value and guidelines]. J Radiol. 2004 May;85(5 Pt 2):680-9. doi: 10.1016/s0221-0363(04)97649-4. French. PMID 15238869
- [Result] Tranquart F, Correas JM, Ladam Marcus V, Manzoni P, Vilgrain V, Aube C, Elmaleh A, Chami L, Claudon M, Cuilleron M, Diris B, Garibaldi F, Lucidarme O, Marion D, Beziat C, Rode A, Tasu JP, Trillaud H, Bleuzen A, Le Gouge A, Giraudeau B, Rusch E. [Real-time contrast-enhanced ultrasound in the evaluation of focal liver lesions: diagnostic efficacy and economical issues from a French multicentric study]. J Radiol. 2009 Jan;90(1 Pt 2):109-22. doi: 10.1016/s0221-0363(09)70089-7. French. PMID 19212279